CLINICAL TRIAL: NCT04357860
Title: Clinical Trial of Sarilumab in Adults Hospitalized With COVID-19 Presenting Cytokine Release Syndrome
Brief Title: Clinical Trial of Sarilumab in Adults With COVID-19
Acronym: SARICOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Junta de Andalucia (Other Government); Red Andaluza de Ensayos Clínicos en Enfermedades Infecciosas (Red ANCRAID) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARICOR
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2020-04

CONDITIONS: SARS-CoV 2; SARS
MeSH Terms: interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sarilumab 200 mg (Experimental): Subjects treated with the best available treatment up to 14 days plus Sarilumab 200 mg single dose.
  Interventions: Drug: Sarilumab 200 MG/1.14 ML Subcutaneous Solution [KEVZARA]
- Sarilumab 400 mg (Experimental): Subjects treated with the best available treatment up to 14 days plus Sarilumab 400 mg single dose.
  Interventions: Drug: Sarilumab 400 MG/2.28 ML Subcutaneous Solution [KEVZARA]
- Control (Active Comparator): Subjects treated with the best available treatment up to 14 days.
  Interventions: Drug: Best available treatment

INTERVENTIONS:
Drug: Sarilumab 200 MG/1.14 ML Subcutaneous Solution [KEVZARA] — Best available treatment up to 14 days plus Sarilumab 200 mg
  Arms: Sarilumab 200 mg
Drug: Sarilumab 400 MG/2.28 ML Subcutaneous Solution [KEVZARA] — Best available treatment up to 14 days plus Sarilumab 400 mg
  Arms: Sarilumab 400 mg
Drug: Best available treatment — Best available treatment up to 14 days
  Arms: Control

SUMMARY:
Early administration of sarilumab in hospitalized patients infected with COVID-19 who have pulmonary infiltrates and are at high risk of unfavorable evolution could decrease/prevent progression to acute respiratory distress syndrome (ARDS) requiring high flow nasal oxygenation (HFNO) or either invasive or non-invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and <75 years
* Admission for confirmed respiratory symptoms to COVID-19 based on a positive PCR in a sample of the respiratory tract in the local laboratory in the absence of respiratory distress syndrome requiring ONAF or mechanical ventilation
* Interstitial pneumonia confirmed by chest radiography or CT
* IL-6 levels> 40 pg / ml. In its absence, D-Dimer (DD)> 1500 or> 1000 may be included if progressive increases are documented
* Negative pregnancy test in women of childbearing age
* Signature of informed consent

Exclusion Criteria:

* SOFA score> 6 points
* Patient who, in the researcher's opinion, is not a subsidiary of invasive mechanical ventilation
* Neutrophil count <2 x 103 / μL
* Platelet count <100 x 103 / μL
* ALT or AST levels> 5 times the upper limit of normal
* Severe renal failure (CrCr <30 ml / min)
* Active bacterial infectious process
* Active tuberculosis, history of not completing treatment against tuberculosis, suspicion of extrapulmonary tuberculosis
* History of intestinal ulcer or diverticulitis
* History of hypersensitivity reactions to Sarilumab or its excipients
* Treatment with TNF antagonists
* Previous treatment with anti-IL6 in the previous 30 days
* Chronic prior treatment with corticosteroids at doses greater than 0.5 mg / kg / day of prednisone or equivalent. Yes, inhaled and topical corticosteroids are acceptable
* Concomitant treatment with immunomodulators, among which are Vitamin D or statins. Macrolides such as azithromycin are acceptable
* Patients on immunosuppressive treatment for any cause
* HIV-infected patients with CD4 <200 / mm3
* Past or current history of autoimmune disease or systemic inflammatory disease
* Patients who have received or are planning therapy with immunomodulatory antibodies, including immunoglobulins
* Participation in any clinical trial that evaluated any investigational product in the last 3 months or less than 5 half-lives of the investigational product
* Pregnancy
* Any other condition that, in clinical judgment, prevents adherence to the patient's protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Ventilation requirements | At day 28 or when the subject is discharged (whichever occurs first)
  Proportion of patients requiring or time (in days) until required:
  * High flow nasal oxygenation (HFNO)
  * Non-invasive mechanical ventilation type BiPAP
  * Non-invasive mechanical ventilation type CPAP
  * Invasive mechanical ventilation

SECONDARY OUTCOMES:
Crude mortality | At day 28 or when the subject is discharged (whichever occurs first)
  Crude mortality at 28 days
Time to clinical improvement | At day 28 or when the subject is discharged (whichever occurs first)
  Time to clinical improvement: defined as the mean change or time in days from randomization to any of the following criteria: (i) improvement of two points on the ordinal scale of 7 points of severity or, (ii) hospital discharge with lifetime. The criteria reached before are used. The 7 point gravity scale includes the following categories:
  1. - Not hospitalized with normal activity
  2. - Not hospitalized but unable to have normal activity
  3. - Hospitalized, without requiring oxygen supplementation
  4. - Hospitalized, requiring oxygen supplementation
  5. - Hospitalized, requiring ONAF, non-invasive mechanical ventilation or both
  6. - Hospitalized requiring ECMO, invasive mechanical ventilation or both
  7. - Death
Time until improvement in oxygenation | At day 28 or when the subject is discharged (whichever occurs first)
  Time (in days) until improvement in oxygenation for at least 48 hours:
  * Time to verify an increase in the SpO2 / FiO2 ratio with respect to the worst SpO2 / FiO2 prior to treatment with Sarilumab and stratified according to levels of IL-6 or DD
  * Time to absence of oxygen requirement to maintain saturation in ambient air ≥ 93%
  * Number of days in need of supplemental oxygen
Proportion of patients requiring invasive mechanical ventilation | At day 28 or when the subject is discharged (whichever occurs first)
  Proportion of patients requiring invasive mechanical ventilation in the trial
Proportion of patients having negative COVID-19 CRP at each visit | At day 28 or when the subject is discharged (whichever occurs first)
  Proportion of patients having negative COVID-19 CRP at each visit of the trial
Mean of serum cytokine levels | At day 28 or when the subject is discharged (whichever occurs first)
  Mean of serum cytokine levels: the panel of cytokines to quantify; IL1-��, IL1-β, IL6, IL8, IL10, IL12, IL18, IL38, INFɣ, TNF��, CCL2, CCL3, CCL4, MIF and PAI-1
Adverse events related to medication and its administration | At day 28 or when the subject is discharged (whichever occurs first)
  Incidence of adverse events related to medication and its administration
Incidence in the appearance of serious bacterial, fungal or opportunistic infections | At day 28 or when the subject is discharged (whichever occurs first)
  Incidence in the appearance of serious bacterial, fungal or opportunistic infections in the subjects
Incidence of perforation of the gastrointestinal tract | At day 28 or when the subject is discharged (whichever occurs first)
  Incidence of perforation of the gastrointestinal tract in subjects
Leukocyte and neutrophil count | At day 28 or when the subject is discharged (whichever occurs first)
  Leukocyte and neutrophil count mean
Hemoglobin levels | At day 28 or when the subject is discharged (whichever occurs first)
  Mean hemoglobin levels
Platelet count | At day 28 or when the subject is discharged (whichever occurs first)
  Platelet count mean
Levels of creatinemia | At day 28 or when the subject is discharged (whichever occurs first)
  Average levels of creatinemia
Bilirubin levels | At day 28 or when the subject is discharged (whichever occurs first)
  Average bilirubin levels
ALT and AST levels | At day 28 or when the subject is discharged (whichever occurs first)
  ALT and AST average levels

CONTACTS AND LOCATIONS:
Overall Officials: Julián de la Torre Cisneros, MD, Study Director — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
All the information will be published and it will be available in open access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the end of the trial.
Access Criteria: Contact uicec@imibic.org

REFERENCES:
- [Derived] Merchante N, Carcel S, Garrido-Gracia JC, Trigo-Rodriguez M, Moreno MAE, Leon-Lopez R, Espindola-Gomez R, Alonso EA, Garcia DV, Romero-Palacios A, Perez-Camacho I, Gutierrez-Gutierrez B, Martinez-Marcos FJ, Fernandez-Roldan C, Perez-Crespo PMM, Cano AA, Leon E, Corzo JE, de la Fuente C, Torre-Cisneros J. Early Use of Sarilumab in Patients Hospitalized with COVID-19 Pneumonia and Features of Systemic Inflammation: the SARICOR Randomized Clinical Trial. Antimicrob Agents Chemother. 2022 Feb 15;66(2):e0210721. doi: 10.1128/AAC.02107-21. Epub 2021 Dec 13. PMID 34902262
- [Derived] Leon Lopez R, Fernandez SC, Limia Perez L, Romero Palacios A, Fernandez-Roldan MC, Aguilar Alonso E, Perez Camacho I, Rodriguez-Bano J, Merchante N, Olalla J, Esteban-Moreno MA, Santos M, Luque-Pineda A, Torre-Cisneros J. Efficacy and safety of early treatment with sarilumab in hospitalised adults with COVID-19 presenting cytokine release syndrome (SARICOR STUDY): protocol of a phase II, open-label, randomised, multicentre, controlled clinical trial. BMJ Open. 2020 Nov 14;10(11):e039951. doi: 10.1136/bmjopen-2020-039951. PMID 33191263